CLINICAL TRIAL: NCT01464359
Title: T-Cell Depleted Double UCB With Post Transplant IL-2 for Refractory Myeloid Leukemia
Brief Title: T-Cell Depleted Double UCB for Refractory AML
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Masonic Cancer Center, University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MT2011-15
Record Dates: First submitted 2011-11-01; First posted 2011-11-03 (Estimated); Results first posted 2015-05-15 (Estimated); Last update posted 2017-12-28 (Actual); Status verified 2017-12

CONDITIONS: Acute Myelogenous Leukemia; Refractory Acute Myelogenous Leukemia
Keywords: umbilical cord blood transplant
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Allopurinol; fludarabine; fludarabine phosphate; Whole-Body Irradiation; Radiation; Cyclophosphamide; Levetiracetam; Busulfan; Cord Blood Stem Cell Transplantation; Interleukin-2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Patients with Acute Myelogenous Leukemia (Experimental): Patients with chemotherapy refractory Acute Myelogenous Leukemia (AML) after a double T-cell depleted (TCD) umbilical cord blood (UCB) transplantation where the smaller unit is activated overnight in interleukin-2 (IL-2). IL-2 will be given three times weekly for 6 doses beginning on days+3 and days +60 to expand UCB-derived natural killer (NK) cells in vivo.
  Interventions: Drug: Allopurinol; Drug: Fludarabine; Radiation: Total body irradiation; Drug: Cyclophosphamide; Drug: Levetiracetam; Drug: Busulfan; Biological: Umbilical Cord Blood Transplantation; Biological: Interleukin-2

INTERVENTIONS:
Drug: Allopurinol — On Day 8 pre-transplant, start hydration with allopurinol per standard of care.
  Other Names: Zyloprim
Drug: Fludarabine — On Days 7, 6 and 5 pre-transplant, 25 mg/m^2 intravenously over 1 hour.
  Other Names: Fludara
Radiation: Total body irradiation — On Days 5, 4, 3, and 2 pre-transplant, 165 cGy times 2 (330 cGy daily, 1320 total dose) according to the University Of Minnesota Blood and Marrow Transplant Program total body irradiation (TBI) guidelines.
  Other Names: Radiation
Drug: Cyclophosphamide — On Days 7 and 6 pre-transplant, 60 mg/kg intravenously (IV) over 2 hours with a high volume fluid flush and mesna per institutional guidelines.
  Alternate Preparative Therapy For Patients Not Able To Receive TBI: Days 5, 4, 3 and 2 pre-transplant; 50 mg/kg/day IV over 2 hours.
  Other Names: Cytoxan
Drug: Levetiracetam — Alternate Preparative Therapy for Patients Not Able to Receive Total Body Irradiation (TBI): Hydration therapy on Day 10 pre-transplant.
  Other Names: Keppra
Drug: Busulfan — Alternate Preparative Therapy For Patients Not Able To Receive TBI: Days 9, 8, 7 and 6 pre-transplant; 0.8 mg/kg (1.1 mg/kg if <12 kg) intravenously every 6 hours
  Other Names: Myleran
Biological: Umbilical Cord Blood Transplantation — Day 0: Two UCB units will compose the graft. The infusion of the first UCB unit should begin within 15 minutes, and no later than 30 minutes after arrival on the Unit. The UCB unit without IL-2 activation will be infused first, followed by the IL-2 activated unit. Both cords will be infused within 30-60 minutes of each other as deemed clinically safe by the BMT attending.
  Other Names: UCBT
Biological: Interleukin-2 — First Course of IL-2 (begin day +3) post-transplant: For patients ≥ 45 kg, IL-2 will be given at 9 million units every other day for a total of 6 doses subcutaneously. Patients weighing less than 45 kilograms, the IL-2 will be dosed at 5 million units/m^2 every other day for a total of 6 doses.
  Second Course of IL-2 (day +60):
  Patients will receive a second course of IL-2 beginning on Day +60 post transplant to expand and educate the NK cells derived from the UCB graft source.
  Other Names: IL-2

SUMMARY:
This trial is proposes to build on our experience and is designed to maximize early (day 3-14) and late (day 60-71) donor-derived natural killer (NK) cell expansion and function in vivo. The proposed platform will allow us the unique opportunity to compare in vivo function from a transplanted umbilical cord blood (UCB) source (presumed to contain NK progenitors requiring "education" in the recipient).

DETAILED DESCRIPTION:
This single center study will determine the feasibility and safety of using a myeloablative conditioning regimen followed (on day 0) by transplantation with double T-cell depleted (TCD) umbilical cord blood (UCB) units where the unit with fewer mononuclear cells (MNCs)/kg will be selected for overnight IL-2 activation prior to infusion. Beginning on day +3, post transplant IL-2 will be administered thrice weekly, not on consecutive days, for a total of 6 doses to expand UCB derived progenitor cells. Post transplant immune suppression prophylaxis will not be administered with the intent to lessen toxicity and allow allogeneic NK cells to function longer providing better anti-leukemic therapy. However if either UCB unit has more than 5% T-cells, the patient will not receive either course of IL-2. Beginning on day +60 after transplantation, a second course of IL-2 will be administered thrice weekly, not on consecutive days, for a total of 6 doses with the purpose of enhancing the in vivo expansion and education of NK cells derived from engrafting UCB cells.

ELIGIBILITY:
Inclusion Criteria:

* Aged 2 to 45 years with acute myeloid leukemia (AML) who meet one of the following criteria:

  * Primary induction failure defined as no complete remission (CR) after two or three induction cycles (no blast limit).
  * Relapsed AML with low disease burden: For patients >21 through 45 years of age: must have <30% marrow blasts within 14 days of enrollment and be at least 28 days from the start of last therapy. For patients 2 through ≤ 21 years of age: must have >5% marrow blasts after no more than 3 induction attempts.

Patients with prior central nervous system (CNS) involvement are eligible provided that it has been treated and is in remission. CNS therapy (chemotherapy or radiation) should continue as medically indicated during the protocol.

* Have acceptable organ function within 14 days of study registration defined as:

  * Renal: creatinine ≤ 2.0 mg/dL (adult patients) or calculated creatinine clearance > 40 ml/min (pediatric patients)
  * Hepatic: bilirubin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP) ≤ 5 times upper limit of normal
  * Pulmonary function: diffusing lung capacity for carbon monoxide corrected for hemoglobin (DLCOcorr) > 50% of normal, (oxygen saturation [>92%] can be used in child where pulmonary function tests (PFT's) cannot be obtained)
  * Cardiac: left ventricular ejection fraction ≥ 45%
* Karnofsky Performance Status ≥ 70% (≥ 16 years) or Lansky Play Score ≥ 50 (pediatrics < 16 years)
* Women of childbearing potential must agree to use adequate contraception (diaphragm, birth control pills, injections, intrauterine device [IUD], surgical sterilization, subcutaneous implants, or abstinence, etc.) for the duration of treatment.
* All patients will be questioned about prior exposure to antibody therapy (including OKT3, rituximab, trastuzumab, and gemtuzumab) without affect to eligibility. Patients with prior exposure will have a blood sample collected for human antimouse antibody (HAMA). For patients with no prior antibody therapy exposure, no further action will be taken.
* Voluntary written consent

Exclusion Criteria:

* Active infection at time of enrollment or documented fungal infection within 3 months unless clearance from Infectious Disease
* Evidence of HIV infection or known HIV positive serology
* Pregnant or breast feeding.
* If < or = 21 years old, prior myeloablative transplant within the last 6 months. If > 21 years old prior myeloablative allotransplant or autologous transplant - if prior conditioning regimen included total body irradiation (TBI), then busulfan/cyclophosphamide(BU/CY) prep should be used
* If > 21 years old - extensive prior therapy including > 12 months of any alkylator chemotherapy (etoposide >100 mg/m^2 x 5 days, cyclophosphamide >1 gm/m^2 or mitoxantrone >8 gm/m^2) delivered at 3-4 week intervals or > 6 months alkylator therapy (as above) with extensive radiation (determined by Radiation Oncology, e.g. mantle irradiation for Hodgkin's) and/or prior radiation therapy that makes a patient ineligible for TBI.
* Known hypersensitivity to any of the study agents

Ages: 2 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2011-10; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Verneris, M.D., Principal Investigator — Masonic Cancer Center, University of Minnesota
Locations (1):
- Masonic Cancer Center, University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Patients With Acute Myelogenous Leukemia: Allopurinol: start on Day -8 per institutional guidelines Fludarabine: give on Days -7, -6 and -5, 25 mg/m^2 intravenously (IV) Cyclophosphamide: give on Days -7 and -6, 60 mg/kg IV along with mesna per institutional guidelines Total body irradiation: give on Days -5, -4, -3, and -2, 165 cGy twice daily Double T-cell depleted umbilical cord blood transplantation with activation of one of the units in interleukin-2 (IL-2): give on Day 0 IL-2: start on Day +3 and Day +60, 9 MU subcutaneously three times weekly for 6 doses
  Alternate preparative therapy for patients not able to receive additional radiation
  Levetiracetam (Keppra): begin on Day -10 per institutional guidelines Busulfan: give Day -9 through Day -6, 0.8 mg/kg (1.1 mg/kg if <12 kg) IV every 6 hours Cyclophosphamide: give Day -5 through Day -2, 50 mg/kg/day IV along with mesna per institutional guidelines
Period: Overall Study
Arm/Group | Patients With Acute Myelogenous Leukemia
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Patients With Acute Myelogenous Leukemia
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Disease Free Survival
Description: The primary endpoint is a disease free survival at 3 months in patients with chemotherapy refractory AML after a double T-cell depleted (TCD) umbilical cord blood (UCB) transplantation where one TCD unit is activated overnight in IL-2 followed by the administration of two courses of IL-2 three times a week for 6 doses beginning on day +3 and on day +60 to expand UCB-derived NK cells in vivo.
Time Frame: At 3 months
Measure: Number; unit: participants
Arm/Group | Patients With Acute Myelogenous Leukemia
Number analyzed (Participants) | 3
participants | 1

2. Secondary Outcome: Incidence of Graft Failure
Description: Incidence of graft failure defined as an absolute neutrophil count of less than 500/uL and a bone marrow that is less than 5% cellular (marrow aplasia)
Time Frame: Day 42
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Acute Myelogenous Leukemia
Number analyzed (Participants) | 3
Participants | 0

3. Secondary Outcome: Incidence of Acute Graft-Versus-Host Disease
Time Frame: Day 60
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Acute Myelogenous Leukemia
Number analyzed (Participants) | 3
Participants | 0

4. Secondary Outcome: Transplant-Related Mortality
Time Frame: Day 180 after Transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Acute Myelogenous Leukemia
Number analyzed (Participants) | 3
Participants | 0

5. Secondary Outcome: Clinical Disease Response
Description: Defined as leukemia clearance and complete remission. Patients will be followed for disease response for 1 year from transplantation unless: consent is withdrawal, patient is unevaluable - if a patient is not evaluable, follow only until the resolution or stabilization of treatment related toxicity, new anti-cancer treatment is started, patient is discharged to hospice (terminal) care.
Time Frame: 1 Year from Transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Acute Myelogenous Leukemia
Number analyzed (Participants) | 3
Participants | 2

6. Secondary Outcome: Duration of Survival
Time Frame: 6 months after Transplantation.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Acute Myelogenous Leukemia
Number analyzed (Participants) | 3
Participants | 1

7. Secondary Outcome: Duration of Survival
Time Frame: 1 year after Transplantation.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Acute Myelogenous Leukemia
Number analyzed (Participants) | 3
Participants | 0

8. Secondary Outcome: Duration of Survival
Time Frame: 2 years after Transplantation.
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Acute Myelogenous Leukemia
Number analyzed (Participants) | 3
Participants | 0

9. Secondary Outcome: Clinical Disease Response
Description: Defined as leukemia clearance and complete remission. Patients will be followed for disease response for 2 years from transplantation unless: consent is withdrawal, patient is unevaluable - if a patient is not evaluable, follow only untilthe resolution or stabilization of treatment related toxicity, new anti-cancer treatment is started, patient is discharged to hospice (terminal) care.
Time Frame: 2 Years from Transplantation
Measure: Count of Participants; unit: Participants
Arm/Group | Patients With Acute Myelogenous Leukemia
Number analyzed (Participants) | 3
Participants | 2

ADVERSE EVENTS:
Arm/Group | Patients With Acute Myelogenous Leukemia
Serious Adverse Events (participants affected / at risk) | 2/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Acute Myelogenous Leukemia (N=3)
Infections and infestations - Other, blood culture w/gram positive cocci and CMV (Infections and infestations) | 1
fever (General disorders) | 1
hepatobilliary disorders - Other, veno occlusive disease (Hepatobiliary disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Patients With Acute Myelogenous Leukemia (N=3)
febrile neutropenia (Blood and lymphatic system disorders) | 3
chills (General disorders) | 3
injection site reaction (General disorders) | 2
cholecystitis (Hepatobiliary disorders) | 1
bruising (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
pain of skin (Skin and subcutaneous tissue disorders) | 1
other, rash (Skin and subcutaneous tissue disorders) | 2
Hypertension (Vascular disorders) | 3
Hypotension (Vascular disorders) | 1
other, veno occlusive disease (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No